CLINICAL TRIAL: NCT03021720
Title: Satisfaction of Patients With Trans-Arterial Radial Access: Quality of Life in Uterine Fibroid Embolization Trial
Acronym: SPARQLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, John Kachura, Interventional Radiologist; Associate Professor of Medical Imaging, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16-0227-A
Record Dates: First submitted 2017-01-09; First posted 2017-01-16 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Uterine Fibroid
Keywords: Uterine fibroid embolization; Uterine artery embolization; Arterial access; Radial access; Interventional radiology; Quality of life; Patient Satisfaction; Patient centered care; Uterine fibroid
MeSH Terms: conditions — Leiomyoma; Patient Satisfaction | interventions — Vascular Access Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral arterial access (Active Comparator): Femoral arterial puncture for the uterine fibroid embolization procedure
  Interventions: Procedure: Arterial access
- Radial arterial access (Experimental): Radial arterial puncture for the uterine fibroid embolization procedure
  Interventions: Procedure: Arterial access

INTERVENTIONS:
Procedure: Arterial access — Location of arterial puncture

SUMMARY:
Randomized trial comparing uterine fibroid embolization patient satisfaction and quality of life with femoral versus radial arterial access

DETAILED DESCRIPTION:
1:1 randomized trial comparing patient satisfaction and quality of life with femoral versus radial arterial access for uterine fibroid embolization

ELIGIBILITY:
Inclusion Criteria:

* Meeting standard eligibility criteria for uterine fibroid embolization
* Satisfactory ulnopalmar arch patency

Exclusion Criteria:

* Unable to provide informed consent
* Unable or unwilling to complete the study questionnaires
* Failed Barbeau test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | From date of procedure to one month after procedure
  Based on visual analog scale (min 0, max 10; higher score indicates better outcome)

SECONDARY OUTCOMES:
Procedure related complication rate | Up to one month after procedure
  Complications categorized based on the Society of Interventional Radiology Standards of Practice Guideline
Procedure time | Duration of intra-procedural time
  Procedure time
Fluoroscopy Time | Duration of intra-procedural fluoroscopy
  Fluoroscopy time used during the procedure
Procedure equipment cost | Procedure
  Cost of disposable equipment used for the procedure
Health related quality of life | 1 month post procedure
  Health related quality of life short form-8 questionnaire (raw score converted to standardised score min 0, max 100; higher score indicates better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: John Kachura, Principal Investigator — Mount Sinai Hospital, University Health Network
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No